CLINICAL TRIAL: NCT04786561
Title: Depression as Risk Factor for Dementia
Brief Title: Depression, Anxiety and Social Relationships as Risk Factors for Dementia
Status: Completed | Type: Observational
Sponsor: Norwegian Centre for Ageing and Health (Other)
Collaborators: Norwegian Health Association (Other); Norwegian University of Science and Technology (Other); Norwegian Institute of Public Health (Other Government); University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 181011
Record Dates: First submitted 2020-02-06; First posted 2021-03-08 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Dementia; Dementia Alzheimers; Risk Factor; Depression; Anxiety; Social Isolation; Loneliness
MeSH Terms: conditions — Dementia; Alzheimer Disease; Depression; Anxiety Disorders; Social Isolation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HUNT4 70+: All inhabitants of Nord-Trøndelag 70 years or older were invited to participate in HUNT 4 70+. HUNT4 refers to the fourth wave of the HUNT-study (HelseUndersøkelse i Nord-Trøndelag or health survey in northern part of Trøndelag community in Middle of Norway) and 70+ refers to the part of the survey directed to participants aged seventy years and older.
- HUNT4 70+ Trondheim: All inhabitants of one district in Trondheim 70 years or older were invited to participate in HUNT 4 70+

SUMMARY:
The main objective of the present work is to establish a firm knowledge base regarding depression and anxiety as risk factors for dementia and how social relationships impact this association. This risk factors, and efforts to reduce them are described through a follow up over three decades.

DETAILED DESCRIPTION:
The Health Study in Nord-Trondelag (HUNT) fulfils most of the key requirements of a population-representative cohort study by meeting the following elements: firm knowledge about the population denominator, knowledge about reasons for refusal (in line with previous methods in HUNT), options for levels and localisation of participation (at test station, at home, at nursing homes), coverage of sociodemographic features by the comprehensive HUNT4-protocol and register linkage, inclusion of institutionalized individuals and individuals with reduced capacity to consent, measurement of risk and compensatory factors across the life course by merging with previous results in HUNT surveys and linkage to registries, core elements and assessment methods can be compared with other European populations studies including elderly people, and finally, the ability to include biobank results in the data analysis. The HUNT data supplemented by register linkage include all established and suspected risk factors of dementia.

A particular focus on primary health care is appropriate because it is in this part of the health care system that the need for extra resources due to the substantial increase in dementia prevalence is most pronounced. Furthermore, preventive measures in a life-course perspective will mainly have to be implemented in the primary health care setting.

ELIGIBILITY:
Inclusion Criteria:

* Living in designated area

Exclusion Criteria:

* None

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Inhabitants living in the designated areas that voluntared to the health survey and accepted a cognitive test.
Sampling Method: Non-Probability Sample
Enrollment: 11000 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of dementia diagnosis in HUNT4 70+ study | 2017-2019
  Two clinical and scientific experts will independently set at diagnosis of cognitive impairment or dementia based on all available information applying standard diagnostic criteria DSM-5.
Incidence of Minimal Cognitive Impairment (MCI) in the HUNT 70+ study | 2017-2019
  Two clinical and scientific experts will independently set at diagnosis of cognitive impairment or dementia based on all available information applying standard diagnostic criteria DSM-5.

SECONDARY OUTCOMES:
Change in loneliness | 1995-2019
  Self-reported feeling of loneliness

CONTACTS AND LOCATIONS:
Overall Officials: Geir Selbæk, Phd, Principal Investigator — Norwegian National Advisory Unit on Ageing and Health
Locations (1):
- Norwegian national advisory unit on Ageing and Health, Tønsberg, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aunsmo RH, Strand BH, Bergh S, Hansen T, Kivimaki M, Kohler S, Krokstad S, Langballe EM, Livingston G, Matthews FE, Selbaek G. Loneliness trajectories and dementia risk: Insights from the HUNT cohort study. Alzheimers Dement (Amst). 2025 Jul 29;17(3):e70154. doi: 10.1002/dad2.70154. eCollection 2025 Jul-Sep. PMID 40735047